CLINICAL TRIAL: NCT06229392
Title: A Phase I Study to Evaluate the Intratumoral Influenza Vaccine Administration in Patients With Breast Cancer
Brief Title: A Study to Evaluate the Intratumoral Influenza Vaccine Administration in Patients With Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Ruta Rao, Study Principal Investigator, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21083002
Record Dates: First submitted 2024-01-05; First posted 2024-01-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Breast Cancer Triple Negative
Keywords: Breast cancer; Breast cancer triple negative; Breast cancer HER2+; Flu vaccine; Intratumoral flu vaccine; Intratumoral vaccine
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intratumoral influenza vaccine (Experimental)
  Interventions: Biological: Fluzone Quadrivalent

INTERVENTIONS:
Biological: Fluzone Quadrivalent — Successive cohorts of participants (3 participants per tumor type per cohort) will each be started on a fixed dose of the influenza vaccine. For the first cohort, patients will receive Fluzone Quadrivalent - (Sanofi Pasteur) - 60mcg/0.5mL (standard dose IT flu shot, or dose level 0) intratumorally on day -6 +/- 1 day and day 0 or 1. For the second cohort, patients will receive Fluzone High-Dose Quadrivalent - (Sanofi Pasteur) - 240mcg/0.7mL (high dose IT flu shot, or dose level 1) intratumorally on day -6 +/- 1 day and day 0 or 1. has context menu

SUMMARY:
This Phase 1 study will assess the safety and efficacy (usefulness) of administering 2 doses of seasonal flu vaccine directly into breast cancer tissue (primary tumor), and will study the tumor and whole body response to the vaccine. If the tumor is palpable (able to fee by touch), the vaccine will be administered by a Surgeon/oncologist in the outpatient floor - both experienced and trained. If not palpable, the procedure will be done via guided Ultrasound by our Breast Radiologist -- both experienced and trained. Women with triple-negative (TNBC) and HER2+ types of breast cancer will be eligible for enrollment. Up to 18 subjects may be enrolled at Rush. Successive groups of 3 subjects per breast cancer type will be given increasing doses of vaccine. There are 3 potential dosing groups (half-dose, full dose, and high dose). Blood, stool (optional), and tumor tissue samples will be collected and tested. The active participation period is from one week prior to starting chemotherapy through three months post surgery.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-2
* Patients must be planning to receive standard of car e neoadjuvant chemotherapy as defined by the most recent version of NCCN guidelines (www.nccn.org)
* Patients must have histologically or cytologically confirmed invasive breast cancer that is either triple-negative or HER2+ (regardless of hormone receptor status)

Exclusion Criteria:

* Patients with any uncontrolled intercurrent illness.
* Patients who have any underlying medical condition for which, in the investigator's opinion, participation would not be in the best interest of the participant
* History of egg allergy
* Patients currently on anticoagulant therapy, corticosteroids, or immunosuppressive agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the seasonal flu vaccine.
* History of Guillain-Barré syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose- limiting toxicity (DLT) | 3 months post surgery
  The primary objective of this trial is to assess the safety of intratumoral (IT) influenza vaccine administration in patients with breast cancer receiving neoadjuvant chemotherapy, by evaluating the percentage of patients experiencing dose- limiting toxicity (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Ruta Rao, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT06229392/ICF_000.pdf